CLINICAL TRIAL: NCT06323915
Title: Comparative Study of 3 Multifocal Intraocular Lenses in Murcia
Acronym: C3M
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cristalens Industrie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020_03_C3M
Record Dates: First submitted 2024-03-15; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract | interventions — Lens Implantation, Intraocular; Cataract Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FineVision (Active Comparator): 28 patients will be implanted bilaterally with Intensity FineVision (PhysIOL, Belgium) trifocal IOLs.
  The device is CE-marked and used according to the intended purpose.
  Interventions: Device: intraocular lens implantation in cataract surgery
- Artis Symbiose (Active Comparator): 28 patients will be implanted bilaterally with Artis Symbiose (Cristalens Industrie, France) IOLs.
  The device is CE-marked and used according to the intended purpose.
  Interventions: Device: intraocular lens implantation in cataract surgery
- Synergy (Active Comparator): 28 patients will be implanted bilaterally with Tecnis Synergy model ZFR00V (Johnson & Johnson, USA) IOLs.
  The device is CE-marked and used according to the intended purpose.
  Interventions: Device: intraocular lens implantation in cataract surgery

INTERVENTIONS:
Device: intraocular lens implantation in cataract surgery — Implantation of intra ocular lenses in both patient's eyes in remplacement of the natural cataracted cristallin that has been removed from the patient's eye during the cataract surgery

SUMMARY:
The goal of this clinical trial is to compare the performance of 3 intraocular lenses (IOLs): FineVision (comparator), ARTIS SYMBIOSE (study lenses), and Tecnis Synergy (comparator) through binocular distance-corrected defocus curve.

This main objective will be to show superiority of the ARTIS SYMBIOSE system through binocular distance-corrected defocus curve.

The patient population to be included is patient suffering from cataract who requires cataract surgery procedure that meet the inclusion and non-inclusion criteria and provide written informed consent.

Participants will attend a total of 5 study visits: 1 preoperative visit, 1 surgery visit and 3 postoperative visits.

DETAILED DESCRIPTION:
This trial is a single center, prospective, randomized (1:1), unblinded, controlled study conducted in Spain according to Art. 82 MDR (PMCF study).

The lead investigator at the Murcia Clínica Vista Ircovisión (Murcia Ircovision Eye Clinic) is Dr. Jerónimo LAJARA BLESA.

This study examines the visual performance of the three IOLs involved : ARTIS Symbiose (study lens) compared to FineVision (comparator), and Tecnis Synergy (comparator) in bilaterally implanted patients.

Due to the design of the ARTIS SYMBIOSE set of multifocal IOLs and the Tecnis Synergy multifocal IOL that target continuous sharp vision from far vision to near vision, this comparative trial is needed to evaluate if these approaches are able to achieve the enhancement in the patients' depth-of-field that has been reported with the FineVision trifocal IOL, which is considered as the "gold standard".

A total of approximately 84 patients will be included at 1 clinical center. Subjects participating in the study will attend a maximum of 5 study visits (1 preoperative, 1 operative and 3 postoperative visits) over a period of 12 months.

Only patients who have age-related cataracts will be included in the study. To participate in this study, patients must be at least 50 years old at the time of screening and maximum 85 years old. All patients who would like to take part in this study will receive a detailed study information by the investigator staff and a written informed form. Before a patient is admitted, he or she must sign a consent form.

The primary study endpoint is to compare the performance of 3 IOLs (FineVision, ARTIS SYMBIOSE, and Tecnis Synergy) through binocular distance-corrected defocus curve.

The entire study including data processing will be carried out in accordance with EN ISO 14155:2020 Clinical Investigation of Medical Devices for Human Subjects, EN ISO 11979-7:2018: Clinical investigations of intraocular lenses for the correction of aphakia, EU MDR 2017/745, MEDDEV 2.7.1 rev. 4 Clinical Evaluation: A Guide for Manufacturers and Notified Bodies, MPDG:2020: Medical Device Law Implementation Act, as well as applicable local regulations and the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* 50 < Age < 85 years old
* Bilateral age-related cataract
* Signed informed consent of the study
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Qualify for bilateral implantation within 1 month
* No previous refractive or ocular surgery
* Need for IOL in this diopter range: 10 to 30 D
* Expected postoperative astigmatism ≤ 0.75 D
* Eye dryness ≤ 2 in dry eye severity grading

Non-inclusion criteria:

* Being under guardianship / curatorship
* Illiterate or not enough knowledge of Spanish language
* Acute or chronic disease or illness that would increase risk or confound study results found to be relevant by the investigators
* Pupil > 4mm or < 2mm in photopic conditions
* Occupation requiring night-time driving or any occupation incompatible with multifocality
* Amblyopia, strabismus, color blindness
* Extremely shallow anterior chamber
* Capsule or zonular abnormalities that may affect postoperative centration or tilt of the lens (e.g. pseudoexfoliation syndrome, uveitis, Marfan's syndrome).
* Pupil abnormalities (non-reactive, tonic pupils, abnormally shaped pupils or pupils that do not dilate under mesopic/scotopic conditions).
* Irregular astigmatism, unstable cornea.

Exclusion Criteria:

* Inability to place the intraocular lens safely at the location planned
* Surgical complications (e.g. non-circular rhexis, oversized or undersized rhexis). Each patient with these intraoperative complications should not be implanted with the study IOL

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2025-09-20 (Estimated)

PRIMARY OUTCOMES:
defocus curve comparison | one month
  The defocus curves will be carried out from + 1.00 D to - 4.00D with measures of binocular visual acuity in LogMAR with ETDRS (Early Treatment Diabetic Retinopathy Study) chart at 1 month.
  The primary endpoint is visual acuity assessed by depth of field at 0 logMAR.

CONTACTS AND LOCATIONS:
Locations (1):
- Vista Clinic Ircovision Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No